CLINICAL TRIAL: NCT00937417
Title: Phase I Study of the Pharmacokinetics and Pharmacodynamics of ZD6474 in Combination With Docetaxel in Advanced Solid Tumors
Brief Title: S0716 Vandetanib and Docetaxel in Treating Patients With Advanced Solid Tumors
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Withdrawn because SWOG no longer pursuing this study at this time
Sponsor: SWOG Cancer Research Network (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: S0716; SWOG-S0716
Record Dates: First submitted 2009-07-10; First posted 2009-07-13 (Estimated); Last update posted 2017-04-24 (Actual); Status verified 2017-04

CONDITIONS: Breast Cancer; Head and Neck Cancer; Lung Cancer; Prostate Cancer; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: unspecified adult solid tumor, protocol specific; recurrent non-small cell lung cancer; stage IV non-small cell lung cancer; stage IV breast cancer; recurrent squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the hypopharynx; recurrent squamous cell carcinoma of the larynx; recurrent verrucous carcinoma of the larynx; stage IV squamous cell carcinoma of the larynx; stage IV verrucous carcinoma of the larynx; recurrent adenoid cystic carcinoma of the oral cavity; recurrent mucoepidermoid carcinoma of the oral cavity; recurrent squamous cell carcinoma of the lip and oral cavity; recurrent verrucous carcinoma of the oral cavity; recurrent basal cell carcinoma of the lip; stage IV adenoid cystic carcinoma of the oral cavity; stage IV basal cell carcinoma of the lip; stage IV mucoepidermoid carcinoma of the oral cavity; stage IV squamous cell carcinoma of the lip and oral cavity; stage IV verrucous carcinoma of the oral cavity; recurrent metastatic squamous neck cancer with occult primary; recurrent lymphoepithelioma of the nasopharynx; recurrent squamous cell carcinoma of the nasopharynx; stage IV lymphoepithelioma of the nasopharynx; stage IV squamous cell carcinoma of the nasopharynx; recurrent lymphoepithelioma of the oropharynx; recurrent squamous cell carcinoma of the oropharynx; stage IV lymphoepithelioma of the oropharynx; stage IV squamous cell carcinoma of the oropharynx; recurrent esthesioneuroblastoma of the paranasal sinus and nasal cavity; recurrent inverted papilloma of the paranasal sinus and nasal cavity; recurrent midline lethal granuloma of the paranasal sinus and nasal cavity; recurrent squamous cell carcinoma of the paranasal sinus and nasal cavity; stage IV esthesioneuroblastoma of the paranasal sinus and nasal cavity; stage IV inverted papilloma of the paranasal sinus and nasal cavity; stage IV midline lethal granuloma of the paranasal sinus and nasal cavity; stage IV squamous cell carcinoma of the paranasal sinus and nasal cavity; recurrent salivary gland cancer; stage IV salivary gland cancer; anaplastic thyroid cancer; stage IV follicular thyroid cancer; insular thyroid cancer; stage IV papillary thyroid cancer; recurrent thyroid cancer; thyroid gland medullary carcinoma; recurrent prostate cancer; hormone-resistant prostate cancer; recurrent breast cancer; stage IV prostate cancer; male breast cancer
MeSH Terms: conditions — Breast Neoplasms; Head and Neck Neoplasms; Lung Neoplasms; Prostatic Neoplasms; Carcinoma, Non-Small-Cell Lung; Squamous Cell Carcinoma of Head and Neck; Esthesioneuroblastoma, Olfactory; Salivary Gland Neoplasms; Thyroid Carcinoma, Anaplastic; Adenocarcinoma, Follicular; Thyroid Cancer, Papillary; Thyroid Neoplasms; Carcinoma, Medullary; Breast Neoplasms, Male | interventions — Docetaxel; vandetanib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm 1 (Experimental): vandetanib and docetaxel
  Interventions: Drug: docetaxel; Drug: vandetanib; Genetic: proteomic profiling; Other: laboratory biomarker analysis; Other: pharmacological study

INTERVENTIONS:
Drug: docetaxel
Drug: vandetanib
Genetic: proteomic profiling
Other: laboratory biomarker analysis
Other: pharmacological study

SUMMARY:
RATIONALE: Vandetanib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor. Drugs used in chemotherapy, such as docetaxel, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving vandetanib together with docetaxel may kill more tumor cells.

PURPOSE: This phase I trial is studying the side effects and best dose of vandetanib given together with docetaxel in treating patients with advanced solid tumors.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To investigate the differential biological effects in tumor tissues through pharmacodynamic endpoints (percent inhibition of pERK, pKDR, and pEGFR) and their correlation with pharmacokinetics of vandetanib in combination with docetaxel in patients with advanced solid tumors.
* To correlate the pharmacodynamic endpoints with the pharmacokinetics of this combination regimen in these patients.
* To recommend an optimal biological dose of this combination regimen for further testing.

Secondary

* To correlate the pharmacokinetics with safety profiles of two dose levels of vandetanib when given in combination with docetaxel.
* To investigate scientific correlates, including serum proteomics and microvessel density (CD31) and cell death (TUNEL) using tumor tissue biopsy samples taken at baseline and during treatment.
* To determine the objective response in patients with measurable disease at baseline.

OUTLINE: This is a multicenter study.

Patients receive docetaxel IV over 1 hour on day 1 and oral vandetanib once daily on days 1-21. Courses repeat every 21 days in the absence of disease progression or unacceptable toxicity. After 6 weeks of treatment, patients who experience clinical benefit but poor tolerance to docetaxel may continue treatment with vandetanib alone.

Plasma samples are collected periodically for pharmacokinetic analysis, measurement of vandetanib trough levels, serum biomarker analysis, and serum proteomics. Tumor tissue samples are collected at baseline and once between days 36-38 for pharmacodynamic analysis.

After completion of study treatment, patients are followed up for up to 28 days.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed advanced solid tumor, including, but not limited to the following:

  * Non-small cell lung cancer
  * Metastatic breast cancer
  * Hormone-refractory prostate cancer
  * Locally recurrent or metastatic head and neck cancer (including thyroid origin)
* Disease for which no standard therapy exists
* Tumor amenable to biopsy
* Measurable or non-measurable disease
* Brain metastases allowed provided patient has undergone brain irradiation (whole brain or gamma knife) AND the metastases have been clinically and radiologically stable for ≥ 6 weeks after completion of irradiation

  * Patients requiring corticosteroids or anticonvulsants for brain metastases must be on a stable or decreasing dose of corticosteroids and seizure free for ≥ 28 days before study enrollment

PATIENT CHARACTERISTICS:

* Zubrod performance status 0-1
* ANC ≥ 1,500/mm^3
* Platelet count ≥ 100,000/mm^3
* SGOT or SGPT ≤ 2.5 times upper limit of normal (ULN)
* Bilirubin ≤ 1.5 times ULN
* PT/INR ≤ 1.1 times normal
* Serum creatinine ≤ 1.8 times ULN OR measured or estimated creatinine clearance > 50 mL/min
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for ≥ 3 months after completion of study treatment
* Willing to undergo two tumor biopsies and blood and tissue sample submission for correlative laboratory studies
* No clinically significant cardiovascular event, including any of the following:

  * Myocardial infarction or cerebrovascular accident within the past 3 months
  * Unstable angina pectoris
  * NYHA class II-IV heart disease within the past 3 months
  * Symptomatic congestive heart failure
  * Serious cardiac arrhythmia
* No history of cardiac disease that, in the investigator's opinion, increases the risk of ventricular arrhythmia
* No history of arrhythmia that is symptomatic or requires treatment (CTCAE grade 3), including any of the following:

  * Multifocal premature ventricular contractions (PVCs)
  * Bigeminy or trigeminy
  * Ventricular tachycardia
  * Uncontrolled atrial fibrillation

    * Medically controlled atrial fibrillation allowed
* No asymptomatic sustained ventricular tachycardia
* No history of or evidence of any of the following on ECG:

  * History of QTc prolongation as a result from other medication that required discontinuation of that medication
  * Congenital long QT syndrome
  * First degree relative with unexplained sudden death under 40 years of age
  * Presence of left bundle branch block
  * QTc with Bazett's correction that is unmeasurable or ≥ 480 msec on screening ECG
* No uncontrolled hypertension, defined as consistent systolic BP > 160 mm Hg or consistent diastolic BP > 100 mm Hg despite medical management
* No intractable nausea or vomiting
* No concurrent active diarrhea that may affect the ability to absorb or tolerate vandetanib
* No gastrointestinal (GI) tract disease resulting in malabsorption syndrome or a requirement for IV alimentation
* No uncontrolled inflammatory GI disease (e.g., Crohn's disease or ulcerative colitis)
* No history of allergic reactions attributed to docetaxel or compounds of similar chemical or biological composition to vandetanib, including other quinazoline compounds (e.g., gefitinib or erlotinib)
* No history of deep venous thrombosis or pulmonary embolism requiring therapeutic anticoagulation
* No known HIV positivity
* No other concurrent uncontrolled illness, including, but not limited to the following:

  * Ongoing or serious active infection
  * Psychiatric illness or social situation that would limit compliance with study requirements
* Prior or concurrent malignancies of other histologies within the past 5 years allowed

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Recovered from prior therapy (i.e., ≤ grade 2 alopecia and ≤ grade 1 toxicity from all other adverse events)
* Prior docetaxel as monotherapy or in combination with other chemotherapeutic agents allowed provided there is potential clinical benefit present, in the investigator's opinion, from the combination of docetaxel and vandetanib
* No prior vandetanib
* No prior surgical procedures affecting absorption
* More than 14 days since prior drugs with a short half-life (e.g., sorafenib or sunitinib) (approval by study coordinator required)
* More than 28 days since prior major surgery, chemotherapy, or radiotherapy
* More than 28 days since prior investigational agents
* More than 2 weeks since prior and no concurrent medications associated with a risk of causing Torsades de Pointes
* No concurrent therapeutic anticoagulation (coumadin, warfarin, or low-molecular weight heparin)

  * Low-dose anticoagulation for indwelling catheter maintenance allowed
* No concurrent medication that may cause QTc prolongation
* No other concurrent chemotherapy, hormonal therapy, radiotherapy, immunotherapy, or any other type of therapy for the treatment of cancer, except for the following:

  * Luteinizing hormone-releasing hormone agonists
  * Bisphosphonates

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2008-09; Primary Completion 2009-09 (Estimated); Study Completion 2009-09 (Estimated)

PRIMARY OUTCOMES:
Pharmacodynamic parameters (percent inhibition of pERK, pKDR, and pEGFR) | 6 months

SECONDARY OUTCOMES:
Correlation of pharmacokinetic profile with pharmacodynamic data and treatment-related toxicities | 6 months
Association between scientific correlates (microvessel density, cell death, circulating endothelial cells, ERK and pERK, and serum proteomics) and treatment outcomes and other patient characteristics | 6 months
Objective tumor response and clinically stable disease in patients with measurable disease at baseline | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Monica Mita, MD, Study Chair — Cancer Therapy and Research Center, Texas

IPD SHARING:
Plan to Share IPD: No